CLINICAL TRIAL: NCT04881188
Title: Risk and Protective Factors in Multimodal Pain Therapy in Patients With Chronic Lumbal Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Katholisches Klinikum Bochum (Unknown)
Responsible Party: Principal Investigator, Claudia Levenig, Researcher, Ruhr University of Bochum
Other Study IDs: MST2020
Record Dates: First submitted 2021-04-30; First posted 2021-05-11 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Chronic Low-back Pain
Keywords: multimodal pain therapy
MeSH Terms: interventions — Fertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic low back pain: Patients suffering from chronic low back pain (duration longer than 3 months) undergoing a multimodal pain therapy
  Interventions: Diagnostic Test: Survey

INTERVENTIONS:
Diagnostic Test: Survey — Patients with chronic low back pain in in-patient multimodal pain therapy. Three survey times, questionnaires

SUMMARY:
Results will show important information about potential protective factors which might be relevant for the recovery of patients suffering from low back pain (theoretical basis). On a clinically applied basis we plan the validation of a short screening in concerns of psychosocial risk and protective factors in patients with chronic low back pain undergoing a multimodal pain therapy (MPT), and this for the first time.

Three main aims are: 1. Prospective validation of a short screening on a theoretical basis for the collection of psychosocial risk factors concerning of an unfavourable therapeutic process in MPT. 2. the verification of differences in subgroups with regard to pain management on a basis of the Avoidance Endurance Model in the development of pain and pain-related disability. 3. The evaluation of potential psychosocial protective factors supporting a positive outcome of MPT, such as resilience, acceptance, self-compassion, and body image.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is one of the most common causes of disease-related disabilities with regard to work ability, physical activity, and mobility, as well as in the development of depressive disorders and cognitive impairments. The multimodal pain therapy (MPT) is a multidisciplinary offer of medical, psychlogical and physiotherapeutic treatment. Currently, MPT is the best therapeutic option. However, there are still many non-responders. It is unknown, which patients will benefit from MPT and which contents are the most effective. Besides somatic factors, the relevance of psychosocial risk factors, such as dysfunctional pain management or disstress and depression, are evident in patients suffering from CLBP. Concepts, such as the Avoidance-Endurance Model of pain (AEM) describe different pattern with regard of mood and pain management, offering an individual therapy. Patients with a fear-avoidance response pattern (FAR) and physical inactivity as well as patients with a depressive endurance response pattern (DER) and physical overactiviity show a poorer response to therapeutical and rehabilitative treatments. On the other side, patients with an adaptive response pattern (AR) and moderate physical activity, and patients with an eustress endurance response pattern (EER) react positive to MPT. If the relevance of these pattern will be shown in patients with CLBP, this would stand for a more individualised therapy concerning psychological and physiotherapeutical treatment (e.g., ExposureTherapy, Pacing). Currently it is unknown which factors are relevant for recovery in patients with AR. One possible protective factor is the personality factor "resilience". The current research situation in the field of chronic pain and resilience is still in its early days and raises the question, if partial aspects such as a high degree of pain acceptance, of self-compassion, and a positive body image show more directly and more clearly relations to a positive response to treatment. Furthermore, research has focused on cross-sectional studies. However, only prospective longitudinal studies will provide insight in cause-and-effect-relationship. On a clinically applied basis the diagnosis of risk and protective factors will play an outstanding role to establish a more individualised therapy and rehabilitation, as also the MPT.

For the diagnosis of the different pain pattern postulated by the AEM, the 9-item Avoidance Endurance Fast-Screen (AEFS) is a reliable and valid short screening. However, it has been investigated in patients with acute pain, so far. A separate validation for patients with CLPB is necessary. Our working group wants to tie up the planned prospective study to preliminary work and show for the first time processes of patients with CLBP undergoing MPT.

On a theoretical basis results will be informative about possible protective factors being important for recovery. On a clinically applied basis we plan the validation of a short-screening of psychosocial risk- and protective factors in patients with CLBP undergoing MPT.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain

Exclusion Criteria:

* acute inflammatory diseases
* acute fractures
* pregnancy
* neurological dieases
* psychiatric diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: in-patients pain clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Chronic Pain Score (von Korff) | 15 weeks
  change of pain intensity from baseline to 3-months-follow up (three time points); minimum value 0 (no pain), maximum value 10 (worst pain possible), higher scores mean a worse outcome
Chronic Disability Score (von Korff) | 15 weeks
  change of pain-related disability from baseline to 3-months-follow up (three time points); minimum value 0 (no disability), maximum value 10 (worst disability possible), higher scores mean a worse outcome

SECONDARY OUTCOMES:
Resilience Scale-13 (RS-13) | first day of study participation
  resilience - thinking and action; 7-point-scale (1 I do not agree - 7 I totally agree); higher scores indicate higher levels of resilience
Chronic Pain Acceptance Questionnaire (CPAQ) | first day of study participation
  Acceptance of chronic pain (subscales "pain willingness" and "activity engagement"), 7-point-scale (0 never - 6 always true); higher scores indicate higher levels of acceptance
Self-compassion Scale (SCS) | first day of study participation
  Self-compassion - how individuals typically act towards themself in difficult times; subscales: self-kindness, self-judgement, common humanity, isolation, mindfulness, over-identification; 5-point-scale (1 almost never - 5 almost always); mean score; higher scores indicate higher levels of self-compassion
Frankfurter Körperkonzeptskalen (FKKS, Frankfurt Body Concept Scales) | 15 weeks
  body image - cognitions of health, self-efficacy and self-acceptance (three subscales); 7 point-scale (1 I strongly agree - 6 I strongly disagree); higher scores indicate a more positive body image
Fremantle Back Awareness Questionnaire (FreBAQ) | 15 weeks
  body image - perception of the back; 5-point-scale (0 never feels like that - 4 Always, or most of the time feels like that); higher scores indicate a poor outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tobias L Schulte, Prof., Study Chair — Katholisches Klinikum Bochum
Locations (1):
- Katholisches Klinikum, Klinik Blankenstein, Hattingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided